CLINICAL TRIAL: NCT05960942
Title: Application of Esketamine in Anesthesia of Autism Children Undergoing Colonic Transendoscopic Enteral Tubing
Brief Title: Application of Esketamine in Anesthesia of Autism Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Collaborators: Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: esketamine 2023 N001
Record Dates: First submitted 2023-05-25; First posted 2023-07-27 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-07

CONDITIONS: Autism Spectrum Disorder
Keywords: fecal Microbiota Transplantation; transendoscopic enteral tube; Gut microbiota; anaesthesia
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Esketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- propofol-esketamine (Experimental)
  Interventions: Drug: propofol combined with esketamine
- propofol-sufentanil (Active Comparator)
  Interventions: Drug: propofol-sufentanil

INTERVENTIONS:
Drug: propofol combined with esketamine — In group PE, esketamine was firstly administered at a dose of 0.3 mg.kg-1, followed immediately by propofol with a single intravenous dose of 2.0 mg.kg-1.
  Arms: propofol-esketamine
Drug: propofol-sufentanil — In group PS, sufentanil was administered intravenously at a dose of 0.2 μg.kg-1, then 2.0 mg.kg-1 propofol was intravenously injected.
  Arms: propofol-sufentanil

SUMMARY:
Autism Spectrum Disorder (ASD) is a group of serious neurodevelopmental disorders. Autistic children appear with significant frequency for medical services, lots of which requiring procedural sedation or anaesthesia. Autistic children have often been described as difficult to sedate or anesthetize due to a variety of ASD symptoms. It is a challenging task to provide safe and effective sedation during the procedure of colonic TET for FMT in autism children. The investigators intend to explore an optimum anesthetic regimen for autism children undergoing endoscopic procedures.

DETAILED DESCRIPTION:
Autistic children appear with significant frequency for medical services, lots of which requiring procedural sedation or anaesthesia. The participants have often been described as difficult to sedate or anesthetize due to a variety of ASD symptoms. It is a challenging task to provide safe and effective sedation during the procedure of colonic TET for FMT in autism children. The primary objective was to compare the clinical efficacy and safety of propofol-esketamine (PE) with propofol-sufentanil (PS) for deep sedation in the procedure of colonic TET in ASD children. A secondary objective was to compare adverse events (AEs) and recovery in those children during/after either PE or PS sedation.

ELIGIBILITY:
Inclusion Criteria:

* (1) aged 2-12 years;
* (2) diagnosed with ASD by pediatric psychiatrists in accordance with the criteria in the Fifth Edition of Diagnostic and Statistical Manual of Mental Disorders (DSM-V);
* (3) evaluated as American Society of Anesthesiologists (ASA) physical status I-II;
* (4) scheduled for colonic TET procedure.

Exclusion Criteria:

* (1) oral sedation (premedication) before intravenous catheter placement;
* (2) any contraindication to study medications;
* (3) other circumstances in which the investigator determined that a patient was not suitable for participation in the clinical trial.

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
movement score during the procedure | through study completion, an average of 10 minutes
  (1 = no movement; 2 = semipurposeful allowing continuation of the procedure; 3 = vigorous purposeful movements withholding the procedure)
first movement time | Up to 1 hour after the procedure
  the time from arriving Postanesthesia care unit to first gross limb movement after procedure

SECONDARY OUTCOMES:
degree of emergence agitation | Up to 2 hour after the procedure
  1 = calm; 2 = not calm but could be easily calmed; 3 = not easily calmed, moderately agitated or restless; and 4 = combative, excited, or disoriented, trashing around
time to full recovery | Up to 3 hour after the procedure
  achieve modified Aldrete score of 10 with the vital signs being normal and stable
arterial blood pressure | through study completion, an average of 15 minutes
  arterial blood pressure was measured noninvasively
adverse event | Up to 24 hour after the procedure
  (including hypoxia (SpO2 <93% for >10 seconds) or respiratory depression (apnea >15 seconds), hypotension (mean arterial pressure < 20% from baseline) or bradycardia (heart rate < 60 /min and/or decrease in heart rate > 20% from baseline) were recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Sir Run Run Hospital, Nanjing, China

IPD SHARING:
Plan to Share IPD: Undecided